CLINICAL TRIAL: NCT00241020
Title: Evaluation of the Efficacy of Long-acting Release Octreotide in Patients With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CSMS995BFR04
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; Octreotide
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Octreotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (1):
- Octreotide (Experimental)
  Interventions: Drug: Octreotide

INTERVENTIONS:
Drug: Octreotide

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the most common malignant disease worldwide with an increasing incidence in industrialized countries. For patients with advanced HCC no efficient treatment is currently available. The objective of this study is to assess the efficacy and safety of octreotide in patients with advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* HCC diagnosis :
* histologically or cytologically proven HCC
* or association of the three following criteria:
* cirrhosis
* typical measurable mass (> 3cm, by 2 methods)
* serum alpha-foetoprotein (AFP) ≥500 µg/L
* Cancer Liver Italian Program (CLIP) score : 0 to 3
* Not eligible for specific treatment (surgery, percutaneous ablation or chemo-embolization)

Exclusion Criteria:

* Glycemia > 2.5 g/L or hypoglycemia
* Extra hepatic life-threatening disease
* Serum creatinin> 120 µmol/L
* Prothrombin time < 50 %
* Platelet count < 50.000 /µL
* Symptomatic cholelithiasis
* Non-measurable tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2002-06; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Overall Survival

SECONDARY OUTCOMES:
Objective response
Survival without progression
Digestive bleeding
Renal insufficiency
Quality of life
· Safety

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals